CLINICAL TRIAL: NCT01655472
Title: Prospective Ultrasonographic and Magnetic Resonance Imaging (MRI) Assessment of General and Brain Fetal Development in Offspring of Schizophrenic Patients
Brief Title: Schizophrenia Imaging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: TASMC-11-NR-0192-11-CTIL; 18105 (Other Grant/Funding Number: 2010 NARSAD Young Investigator Award)
Record Dates: First submitted 2012-06-30; First posted 2012-08-01 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Foetal Differences Between Healthy and Schizophernic Parents
Keywords: schizophrenia; imaging
MeSH Terms: conditions — Schizophrenia | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- healthy parents (Active Comparator)
  Interventions: Device: imaging follow up: MRI scan; Device: imaging follow up: Ultrasonographic examination
- schizophrenic parents (Active Comparator)
  Interventions: Device: imaging follow up: MRI scan; Device: imaging follow up: Ultrasonographic examination

INTERVENTIONS:
Device: imaging follow up: MRI scan — .1 Psychiatric interview. 2. Questionnaires 3. Blood samples for triple test: alfa feto protein, HCG, E3 4. A thorough fetal ultrasound examination including anatomic screening on 23-24 weeks of pregnancy. 5. A detailed trans-vaginal neurosonographic multi-planer examination, on 32-34 weeks of pregnancy 6. Fetal MRI scan on 32-34 weeks of pregnancy, 7. Newborn brain transfontanelar ultrasonography ,within 2 months postpartum 8. Newborn medical examination within 2 months postpartum.
  Other Names: 1. MRI 1.5 T & 3.0 T, MR systems, GE 1.5 & 3T Signa HDx MR system, General Electric Medical Technologies; 2. GE MEDICAL SYSTEMS, ULTRASOUND, GE Medical Systems Kretztechnik GmBH & Co OHG
Device: imaging follow up: Ultrasonographic examination

SUMMARY:
Schizophrenia is a common disorder with a lifetime prevalence of about 1%.Genetic studies strongly suggest a genetic component to the inheritance of schizophrenia. Structural neuroimaging studies have provided consistent evidence for brain abnormalities in schizophrenia. The timing of brain abnormalities in schizophrenia has not been determined yet.

The investigators hypothesize that brain structural changes can be detected in neonatal life. The investigators hypothesize that offspring of schizophrenic patients will have higher rates of brain structural changes in the neonatal period. The investigators propose to study early development of fetuses in offspring of patients with schizophrenia. The study is a multi-center prospective trial.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who carry an offspring of a schizophrenia patient: whether the mother, the father or both suffer from schizophrenia.

Exclusion Criteria:

* Alcohol or drug abuse of pregnant woman
* Past history or present occurrence of major neurologic or somatic illness
* Genetic disease
* Other psychiatric disorders other than schizophrenia such as Mental retardation
* Bipolar Disorder and Delusional Disorder

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Brain morphological changes between groups | 2 years
  Both MRI scans and US scans will be compared between the groups, assessing brain morphological and volumetric differences .

CONTACTS AND LOCATIONS:
Overall Officials: Nivi Rotenberg, M.D., Principal Investigator — International Diabetes Federation
Locations (8):
- Israel (8):
  - Abarbanel Mental Health Centre, Bat Yam
  - Beer Yaacov Mental health Centre, Beer Yaakov
  - Shalvata mental health centre, Hod HaSharon
  - Edith Wolfson Medical Centre, Holon
  - Geha mental health centre, Petah Tikva
  - Brill outpatient clinic, Tel Aviv
  - Sourasky Medical Centre, Tel Aviv
  - Chaim Sheba medical centre, Tel Litwinsky